CLINICAL TRIAL: NCT01835418
Title: Bedtime Administration of Amlodipine Versus Lisinopril: a Randomized Trial
Brief Title: Bedtime Administration of Amlodipine Versus Lisinopril
Acronym: BAVLART
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Allina Health System (Other)
Responsible Party: Principal Investigator, David Ingham, Physician, Allina Health System
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 9529148100
Record Dates: First submitted 2013-02-21; First posted 2013-04-19 (Estimated); Last update posted 2013-04-19 (Estimated); Status verified 2013-04

CONDITIONS: Hypertension
Keywords: managed with bedtime administration of lisinopril versus amlodipine
MeSH Terms: conditions — Hypertension | interventions — Amlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lisinopril (Experimental): bedtime administration of lisinopril 20mg
  Interventions: Drug: Amlodipine
- Amlodipine (Experimental): Bedtime administration of amlodipine 5mg
  Interventions: Drug: Amlodipine

INTERVENTIONS:
Drug: Amlodipine — crossover comparison of amlodipine vs lisinopril

SUMMARY:
This study seeks to compare the differences in effectiveness among individual patients treated at for hypertension with bedtime administration of amlodipine versus lisinopril. There will be an analysis of whether one medication was more effective than another and whether specific patient factors could predict who responded better to which one.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 to 80
* Newly diagnosed hypertension based on 24 hour ambulatory blood pressure monitor criteria.
* Minimum Asleep SBP mean of ≥ 120mmHg for inclusion.

Exclusion Criteria:

* Current antihypertensive medication use
* Baseline GFR < 45
* Preexisting macroproteinuria
* Chronic congestive heart failure
* History of CVA
* Diabetes Mellitus
* Pregnancy
* Night-shift work
* Other preexisting contraindication to amlodipine or lisinopril

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-04; Primary Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Change in mean sleep-time systolic blood pressure after addition of a bedtime dose of amlodipine versus lisinopril | 1 year

SECONDARY OUTCOMES:
Changes in mean sleep-time diastolic, awake systolic and diastolic blood pressures, including comparison of % achieving target BP | 1 year
Impact of individual medications on sleep-time blood pressure drop (dipping status) | 1 year
Association of baseline renin levels to sleep-time blood pressure drop | 1 year
Association of baseline renin levels with response to amlodipine versus lisinopril | 1 year
Association of baseline dipping status with response to amlodipine versus lisinopril | 1 year
Association of age and response to amlodipine versus lisinopril | 1 year